CLINICAL TRIAL: NCT02450695
Title: A Randomized Crossed-over Trial Examining Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) in Treatment Refractory Obsessive-Compulsive Disorder.
Brief Title: rTMS in Treatment Refractory Obsessive-Compulsive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were recruited.
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0190
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: rTMS; treatment refractory; treatment resistant; SSRI; clomipramine
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): In rTMS, a device called a "stimulator" provides energy to a "magnetic coil". The coil is a handheld unit that delivers magnetic pulses. The coil is placed against the scalp on the top of your head. Sessions will occur once a day, 5 days/week, for 3 weeks.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): The coil in the sham rTMS phase will be positioned 90 degrees off the scalp, with one wind of the coil touching the scalp. This will ensure that the participant will not be affected by the machine during this time. All other factors will be similar to the active rTMS phase.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS

SUMMARY:
This study will evaluate the effectiveness of rTMS as a potential treatment for refractory OCD in a randomized, crossover design.

DETAILED DESCRIPTION:
The study is a minimum of 7 weeks long. In the first treatment phase (three weeks), participants will be randomly assigned to one of two treatment conditions: active rTMS or sham rTMS. The "sham" rTMS is the inactive form of the treatment where the experience during the sessions will be similar to an active rTMS session, but it will have no medical value. During these 3 weeks, they will attend a session each day for 5 days per week at Mood Disorders Clinic located at St. Joseph's Healthcare. Each of these sessions will be an hour long totalling 15 visits in the first 3 weeks. After every 5 sessions they will be asked to complete the following self-report questionnaires: Baratt Impulsiveness Scale, Hamilton Anxiety Rating Scale and the Hamilton Depression Rating Scale. The clinician-rated: Clinical Global Impression Scale and Yale Brown Obsessive Compulsive Scales will also be completed.

The two treatment phases will be separated by a flexible wash-out of a minimum of one week where participants will not attend any visits.

After this, they will begin the second treatment phase (three weeks) which will be the treatment condition they were not previously assigned to. In other words, individuals previously on the active rTMS treatment will now begin sham rTMS treatment and vice versa. These sessions will be identical to those involved in the first treatment phase, except the treatment condition will be different. Before and after each treatment session they will also be asked a series of questions to rate potential rTMS side effects and complete a cognitive task known as the "Go/no-go task."

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of OCD (DSM 5) according to the MINI
* Y-BOCS score of ≥20
* History of treatment-resistant OCD, established by a trained psychiatrist with extensive expertise in the OCD field. Treatment-resistance will be defined as non-response to at least two SRIs trials (clomipramine, fluoxetine, sertraline, paroxetine, fluvoxamine, citalopram, escitalopram).

Exclusion Criteria:

* Any additional current psychiatric comorbidity, except for mild depressive and anxious symptoms
* A lifetime DSM-5 diagnosis of schizophrenia or other psychotic syndromes, substance dependence or substance abuse, including alcohol, bipolar I or II disorder, mental disorder due to a general medical condition
* Serious suicide risk
* Episodic OCD
* Illness duration less than two years
* Hospitalization in the last 6 months
* Pharmacological treatment changes in the last 3 months
* The inability to receive rTMS because of metallic implants, or history of seizures (personal or family history of seizure in first degree relatives)
* Any major medical disease
* Pregnancy or nursing of an infant
* The inability or refusal to provide informed consent
* Prior TMS exposure (in order to reduce the risk of unblinding).

No psychotherapy and/or pharmacological treatment changes will be allowed during the study period. Pharmacologically treated patients should be on constant medications for at least 2 weeks before entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | 7 Weeks

SECONDARY OUTCOMES:
Barratt Impulsiveness Scale | 7 Weeks
Hamilton Anxiety rating Scale | 7 weeks
Hamilton Depression Rating Scale | 7 Weeks
Clinical Global Impression Scale | 7 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Center, Hamilton, Ontario, Canada